CLINICAL TRIAL: NCT05842161
Title: Treatment Development for Smoking Cessation and Engagement in HIV/TB
Brief Title: South Africa Smoking Cessation and Engagement in HIV/TB Care Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other); University of Cape Town (Other)
Responsible Party: Principal Investigator, Conall O'Cleirigh, Director, Behavioral Medicine/Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P000792; 5R34DA057169-03 (NIH)
Record Dates: First submitted 2023-04-12; First posted 2023-05-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HIV Infections; Tuberculosis; Smoking Cessation
MeSH Terms: conditions — HIV Infections; Tuberculosis; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QUIT-AD (Experimental): An six-session adapted cognitive-behavioral intervention for smoking cessation and treatment adherence. Intervention content will include psychoeducation related to cognitive-behavioral therapy, smoking, TB, and HIV; behavioral activation; distress tolerance; and relapse prevention.
  Interventions: Behavioral: QUIT-AD
- Enhanced Treatment as Usual (ETAU) (Active Comparator): After randomization, participants in the ETAU condition will receive one session of psychoeducation on the HIV- and TB-related health benefits of smoking cessation.
  Interventions: Other: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: QUIT-AD — An adapted, six-session cognitive behavioral therapy intervention for smoking cessation and treatment adherence
  Arms: QUIT-AD
Other: Enhanced Treatment as Usual — Standard treatment for HIV/TB with one session of psychoeducation.
  Arms: Enhanced Treatment as Usual (ETAU)

SUMMARY:
The purpose of this study is to integrate elements from existing interventions developed by our team into a single intervention (QUIT-AD), designed to improve smoking cessation and favorable HIV/TB treatment outcomes among individuals with HIV and/or TB in Cape Town, South Africa. If feasibility, acceptability, and preliminary efficacy are demonstrated, the intervention will be ready for large-scale effectiveness/implementation testing. This program will has the potential to dramatically improve public health by increasing the smoking quit rate and facilitating favorable HIV/TB treatment outcomes among patients with HIV and/or TB in resource limited South African settings.

DETAILED DESCRIPTION:
One of the greatest public health challenges facing South Africa (SA) is tobacco use, which fuels the overlapping epidemics of HIV and pulmonary tuberculosis (TB). Tobacco is the single most preventable cause of death globally, causing more than 7 million deaths per year, with 80% of individuals who use tobacco currently residing in low- and middle-income countries (LMICs). Smoking is an independent risk factor for HIV acquisition, higher viral load, and increased rate of progression to AIDS. Similarly, smoking exacerbates risk for TB and compromises TB treatment,12 increasing TB-related morbidity and mortality. Individuals who smoke are twice as likely to be infected with TB, to transition from latent to active TB, and to die from TB. The prevalence of smoking among people with HIV (PWH) in SA is disproportionately high, as is the prevalence of smoking among people with TB. Among men with HIV in SA, 52% are current smokers, significantly higher than in the general population, whereas 13% of women with HIV report current smoking. Similarly, 56% of patients in SA with active TB currently smoke tobacco, and the prevalence of smoking among individuals with suspected and confirmed TB in Cape Town (63% in men, 44% in women), is much higher than in the general population (35% in men, 10% in women). Together, smoking, HIV, and TB are fueling a dangerous increase in chronic obstructive pulmonary disease, which the World Health Organization (WHO) predicts will become the third most common cause of death globally by 2030, increasing the burden of lung disease in resource-limited settings. Given that the intersecting epidemics of smoking, HIV, and TB pose high risk for poor health outcomes, SA is in urgent need of a smoking cessation intervention that also improves engagement in HIV and TB treatment. This project will leverage components of our previous work to culturally adapt an intervention (QUIT-AD) that improves smoking cessation and HIV/TB treatment adherence specifically tailored for PWH and/or TB in SA. Individuals using tobacco who are (a) living with HIV or (b) initiating TB treatment or (c) living with HIV and initiating TB treatment will be recruited to participate. The study will take place in Khayelitsha, a peri-urban settlement in Cape Town.

Our aims are as follows:

Aim 1: To collect qualitative data that will inform the development of QUIT-AD. We will conduct semistructured interviews with PWH and/or TB who use tobacco (n=25-30) and a focus group with providers or other clinic staff (e.g., adherence counselors, pulmonologists; n=6-8). The patient interviews will identify (1) multi-level barriers (i.e., individual, interpersonal, structural) to smoking cessation and (2) the unique ways in which smoking affects engagement in HIV and TB care. The focus group will explore providers' perspectives on barriers to smoking cessation and treatment engagement and will inform the development of the QUIT-AD protocol.

Aim 2: Specify the QUIT-AD manual and conduct a small open trial (n=5) of the intervention. This open trial will enable us to iteratively refine the intervention, the treatment manual, and the study procedures.

Aim 3a: Assess the feasibility and acceptability of QUIT-AD in a pilot randomized controlled trial compared to enhanced (inclusive of basic adherence counseling and psychoeducation) treatment as usual (n=86, 43 per arm, to ensure 62 completers). Secondary outcomes will be biologically-verified point prevalence abstinence, number of cigarettes smoked, favorable HIV (defined as suppressed viral load), favorable TB treatment outcome (defined as absence of TB symptoms and a negative GeneXpert test or a negative sputum culture), or both at 6 months.

Aim 3b: Conduct individual interviews with providers and clinic administrators to inform future implementation (n=10-15). The provider interviews will explore issues that affected implementation of the intervention in the clinic, including intervention characteristics that will support sustainability.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older
2. Willing and able to provide written informed consent
3. Living with HIV, confirmed via medical record, and on antiretroviral therapy (ART) AND/OR within 1 month of initiating or reinitiating TB treatment; positive GeneXpert test or sputum culture

(5) Daily smoker operationalized as > 5 cigarettes per day, (6) Motivation (> 5/10) to quit smoking or > 24 hour quit past yr

Exclusion Criteria:

1. Habitual use of other tobacco products
2. Current interfering untreated/unstable mental health condition (e.g., psychosis, bipolar dx)
3. Current use of non-study pharmacotherapy for smoking cessation,
4. Cognitive Behavioral Therapy for smoking cessation initiated within the past year,
5. Diagnosed with extra-pulmonary or drug resistant (MDR or XDR) TB based upon chart review

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of intervention | At baseline
  Feasibility of administering the QUIT-AD intervention. Will be will be assessed by (1) interventionist fidelity to the protocol (determined by a review of 20% of session audio recordings to document whether all key session themes were addressed), (2) session attendance, and (3) participant retention at the follow-up assessment
Feasibility of intervention | At treatment sessions
  Feasibility of administering the QUIT-AD intervention. Will be will be assessed by (1) interventionist fidelity to the protocol (determined by a review of 20% of session audio recordings to document whether all key session themes were addressed), (2) session attendance, and (3) participant retention at the follow-up assessment
Feasibility of intervention | 2-Month Follow-Up (2 months post treatment initiation)
  Feasibility of administering the QUIT-AD intervention. Will be will be assessed by (1) interventionist fidelity to the protocol (determined by a review of 20% of session audio recordings to document whether all key session themes were addressed), (2) session attendance, and (3) participant retention at the follow-up assessment
Feasibility of intervention | 6-Month Follow-Up (6 months post treatment initiation)
  Feasibility of administering the QUIT-AD intervention. Will be will be assessed by (1) interventionist fidelity to the protocol (determined by a review of 20% of session audio recordings to document whether all key session themes were addressed), (2) session attendance, and (3) participant retention at the follow-up assessment
Acceptability of intervention | At baseline
  How acceptable participants find the QUIT-AD intervention to be. Will be assessed via a brief questionnaire to be completed after every other treatment session; on a five-point Likert style scale, participants will rate the 7 component constructs of the acceptability of health care interventions framework: affective attitude (i.e., how an individual feels about the intervention), burden, ethicality (i.e., the extent to which the intervention aligns with one's value system), intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy.
Acceptability of intervention | At treatment sessions
  How acceptable participants find the QUIT-AD intervention to be. Will be assessed via a brief questionnaire to be completed after every other treatment session; on a five-point Likert style scale, participants will rate the 7 component constructs of the acceptability of health care interventions framework: affective attitude (i.e., how an individual feels about the intervention), burden, ethicality (i.e., the extent to which the intervention aligns with one's value system), intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy.
Acceptability of intervention | 2-Month Follow-Up (2 months post treatment initiation)
  How acceptable participants find the QUIT-AD intervention to be. Will be assessed via a brief questionnaire to be completed after every other treatment session; on a five-point Likert style scale, participants will rate the 7 component constructs of the acceptability of health care interventions framework: affective attitude (i.e., how an individual feels about the intervention), burden, ethicality (i.e., the extent to which the intervention aligns with one's value system), intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy.
Acceptability of intervention | 6-Month Follow-Up (6 months post treatment initiation)
  How acceptable participants find the QUIT-AD intervention to be. Will be assessed via a brief questionnaire to be completed after every other treatment session; on a five-point Likert style scale, participants will rate the 7 component constructs of the acceptability of health care interventions framework: affective attitude (i.e., how an individual feels about the intervention), burden, ethicality (i.e., the extent to which the intervention aligns with one's value system), intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy.

SECONDARY OUTCOMES:
Short-term point prevalence smoking abstinence | 2-Month Follow-Up (2 months post treatment initiation)
  Biologically verified 7-day point prevalence abstinence (PPA). Using the timeline follow-back method (TLFB), participants will self-report the last time they smoked. TLFB results will be biologically verified with saliva cotinine.
Average number of cigarettes smoked over the past 7 days | At baseline
  Using the timeline follow-back method (TLFB), participants will self-report the number of cigarettes they smoked per day in the past 7 days.
Average number of cigarettes smoked over the past 7 days | At each treatment session
  Using the timeline follow-back method (TLFB), participants will self-report the number of cigarettes they smoked per day in the past 7 days.
Average number of cigarettes smoked over the past 7 days | 2-Month Follow-Up (2 months post treatment initiation)
  Using the timeline follow-back method (TLFB), participants will self-report the number of cigarettes they smoked per day in the past 7 days.
Average number of cigarettes smoked over the past 7 days | 6-Month Follow-Up (6 months post treatment initiation)
  Using the timeline follow-back method (TLFB), participants will self-report the number of cigarettes they smoked per day in the past 7 days.
Favorable HIV/TB treatment outcome | 6-Month Follow-Up (6 months post treatment initiation)
  Favorable outcome defined differently based on a given participant's diagnoses. For participants with HIV alone, favorable treatment outcome will be defined as a VL < 1000. For participants with TB alone, favorable treatment outcome will be defined by the following two criteria: absence of all three TB symptoms (productive cough, fever for more than two weeks, night sweats) determined by study nurse review; and a negative GeneXpert test or a negative sputum culture or smear. For participants with both HIV and TB, favorable treatment outcome will be a combined variable with three levels: failing to meet the definition for either favorable HIV or favorable TB outcome (coded as 0), meeting criteria for either favorable HIV or favorable TB treatment outcome (coded as 1), and meeting the definitions for both favorable HIV and TB treatment outcomes (coded as 2).

OTHER OUTCOMES:
Adherence to HIV/TB treatment | At baseline, six treatment sessions, and 2 follow-up visits - over 6 months
  Adherence to HIV and TB treatment will be assessed via self-report and pharmacy refill count. The self-report measure will assess adherence over a 30-day period. For ART, participants will self-report on their adherence using a 3-item validated scale. For TB treatment, the measure will be informed by TB treatment adherence documentation on patients' adherence register/TB card and adapted from our previous work in HIV medication adherence. Pharmacy refill adherence will be calculated as the mean adherence of all drugs in the combination being prescribed at that time point; from this data, a binary measure will be created, and adherence will be defined as 90% or more of days covered in the specified time period.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Stanton, PhD, Principal Investigator — Boston University
Locations (1):
- University of Cape Town, Rondebosch, South Africa

IPD SHARING:
Plan to Share IPD: No